CLINICAL TRIAL: NCT06494878
Title: The PARTUM (Postpartum Aspirin to Reduce Thromboembolism Undue Morbidity) Trial
Brief Title: The PARTUM Trial: Postpartum Aspirin to Reduce Thromboembolism Undue Morbidity
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB24-0317
Record Dates: First submitted 2024-06-12; First posted 2024-07-10 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Venous Thromboembolism; Postpartum Period; Aspirin; Low Molecular Weight Heparin
Keywords: deep vein thrombosis; pulmonary embolism; postpartum; pregnancy; thrombophilia; cesarean delivery; preeclampsia; small-for-gestational age infant; postpartum hemorrhage; postpartum infection
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Thrombophilia; Pre-Eclampsia; Postpartum Hemorrhage | interventions — Aspirin; Heparin, Low-Molecular-Weight; Dalteparin; Enoxaparin; Nadroparin; Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Experimental): Low-dose aspirin (75-100 mg) once daily for 6 weeks.
  Interventions: Drug: Aspirin
- Low-molecular-weight heparin (Active Comparator): Site-specific low-molecular-weight heparin regimen as prescribed by the treating physician.
  Interventions: Drug: Low-molecular-weight heparin

INTERVENTIONS:
Drug: Aspirin — 75-100 mg taken once daily by mouth.
  Arms: Aspirin
Drug: Low-molecular-weight heparin — Low-molecular-weight heparin injections daily as prescribed by the treating physician.
  Other Names: Dalteparin, Enoxaparin, Nadroparin, Tinzaparin
  Arms: Low-molecular-weight heparin

SUMMARY:
The goal of the PARTUM trial is to determine if taking low-dose aspirin daily for 6 weeks after delivery is similar (non-inferior) to usual care low-molecular-weight heparin injections to prevent venous thromboembolism (VTE: blood clots in the legs or lungs) for postpartum individuals with VTE risk factors.

DETAILED DESCRIPTION:
The PARTUM trial design is a Prospective Randomized Open Blinded End-point (PROBE) non-inferiority trial. Participants with risk factors for venous thromboembolism (VTE) as defined by the inclusion criteria will be identified during pregnancy, labor and delivery, and up to 48 hours after delivery.

Eligible and consenting participants will be randomly assigned to one of two study arms: Low-dose aspirin (75-100mg according to country availability) daily for 42 days post-randomization, or a usual care site-specific low-molecular-weight-heparin (LMWH) regimen with the dose and duration of LMWH determined by the participant's healthcare provider.

Follow-up will occur at 6 weeks and 90 days post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* ONE (or more) First Order Criterion:

  1. Known inherited thrombophilia diagnosed prior to enrolment, regardless of family history of VTE:

     i. Heterozygous factor V Leiden, or ii. Heterozygous prothrombin gene variant, or iii. Protein C deficiency, or iv. Protein S deficiency, and/or
  2. Antepartum immobilization for ≥7 days. Immobilization is defined as bed rest with 90% of waking hours spent in bed at any time during the antepartum period AND/OR

TWO (or more) Second Order Criteria:

1. Pre-pregnancy BMI ≥30 kg/m²
2. Smoking in the current pregnancy or within 3 months prior to pregnancy
3. Previous clinical history of superficial vein thrombosis
4. Preeclampsia
5. Current pregnancy ending in stillbirth (pregnancy loss >20 weeks gestation)
6. Unplanned cesarean delivery (unplanned = not a scheduled cesarean delivery)
7. Small-for-gestational-age infant at time of delivery (<3rd percentile adjusted for gestational age and sex)
8. Peripartum or postpartum infection (symptoms/signs of infection and documented fever and laboratory evidence of infection with positive blood cultures or an elevated white blood cell count based on local laboratory cutoffs)
9. Postpartum hemorrhage (≥1000 mL of blood loss, regardless of delivery mode)

Exclusion Criteria:

1. More than 48 hours since delivery at the time of randomization
2. Received more than 1 dose of LMWH since delivery
3. Need for postpartum LMWH prophylaxis or systemic anticoagulation as judged by their physician and/or local investigator. May include but is not limited to:

   1. Documented history of provoked or unprovoked VTE
   2. Mechanical heart valve(s)
   3. Known antiphospholipid syndrome (APS)
   4. Known high-risk inherited thrombophilia i) Antithrombin deficiency, or ii) Homozygous factor V Leiden, or iii) Homozygous prothrombin gene mutation, or iv) More than 1 thrombophilia: any combination of 2 or more: factor V Leiden, prothrombin gene mutation, protein C deficiency, protein S deficiency
4. Need for postpartum ASA as judged by their physician and/or local investigator. May include but is not limited to:

   1. Documented history of myocardial infarction
   2. Documented history of ischemic stroke or transient ischemic attack (TIA)
5. Active bleeding, excluding normal vaginal bleeding, at the time of randomization
6. Known medical condition as judged by their physician and/or local investigator to be a contraindication to ASA or LMWH including known ASA or LMWH allergy
7. <18 years of age
8. Unable or declined consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8805 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Symptomatic VTE | 6 weeks
  Proximal lower or upper extremity DVT, PE involving segmental or higher arteries or multiple subsegmental arteries, and unusual site [non-limb] venous thromboembolism

SECONDARY OUTCOMES:
Late symptomatic VTE | 90 days
  Proximal lower or upper extremity DVT, PE involving segmental or higher arteries or multiple subsegmental arteries, and unusual site [non-limb] venous thromboembolism
Superficial vein thrombosis | At 6 weeks and at 90 days
  A non-compressible vein segment on ultrasound that involves the superficial veins in the lower or upper extremity
Distal deep vein thrombosis | At 6 weeks and at 90 days
  A non-compressible vein segment on ultrasound involving the deep veins that is distal to the popliteal vein in the lower extremity, or distal to the axillary vein in the upper extremity
Single subsegmental pulmonary embolism (SSPE) | At 6 weeks and at 90 days
  Intraluminal filling defect that involves one subsegmental artery only
Major bleeding | At 6 weeks and at 90 days
  Based on the ISTH definition
Clinically relevant non-major bleeding | At 6 weeks and at 90 days
  Based on the ISTH definition
Wound hematoma requiring intervention | At 6 weeks and at 90 days
  Requiring intervention such as hematoma evacuation or wound packing
Symptomatic arterial thromboembolism | At 6 weeks and at 90 days
  Ischemic stroke/transient ischemic attack, myocardial infarction, or peripheral arterial embolism
Postpartum preeclampsia | At 6 weeks and at 90 days
  New preeclampsia presenting in the postpartum period
Heparin-induced thrombocytopenia | At 6 weeks and at 90 days
  According to a priori categories of definite or possible HIT.
All-cause mortality | At 6 weeks and at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Skeith, MD, Principal Investigator — University of Calgary; Marc Rodger, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (3):
- Canada (3):
  - Foothills Medical Centre, Calgary, Alberta
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request.